CLINICAL TRIAL: NCT04078633
Title: Pilot Studies of Innovative Hand Washing Interventions for Internally Displaced Populations in Ethiopia
Brief Title: Innovative Hand Washing Interventions for Internally Displaced Populations in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Action Contre la Faim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17604
Record Dates: First submitted 2019-08-15; First posted 2019-09-06 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2019-08

CONDITIONS: Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: N/A - the study does not involve drug or biologic products. The study looks at the impact of behavioural interventions
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Normal Liquid Soap (250mL) (Experimental): A normal hygiene kit will be distributed to the households. In addition, a liquid soap will be added to see the impact of having a liquid soap for hand washing on hygiene behaviors.
  Interventions: Behavioral: Hand hygiene interventions
- Bar soap (250gram) (Experimental): A normal hygiene kit will be distributed to the households. In addition, a nice bar soap will be added to see the impact of having a nicer bar soap for hand washing on hygiene behaviors.
  Interventions: Behavioral: Hand hygiene interventions
- Mirror (50x30cm) (Experimental): A normal hygiene kit will be distributed to the households. In addition, a mirror will be added to see the impact of having a mirror by the handwashing stand on handwashing behaviour. The mirror will have a plastic edge and be 30x 50cm in size.
  Interventions: Behavioral: Hand hygiene interventions
- Control (No Intervention): A normal hygiene kit will be distributed to the households. No additional interventions will be given.
- Nurture story for hygiene promotion (Experimental): Hygiene promoters will share a story of being a good parent through teaching their children to do hand washing with soap at critical times. A story about a good mother who every day reminds her child to wash her/his hands before eating or preparing food and after going to the toilet will be shared with participants. The story ends with the child growing up healthy, happy and with a good education. This story if belived to increae handwashing with soap in the household/
  Interventions: Behavioral: Hand hygiene interventions
- Comfort story for hygiene promotion (Experimental): Hygiene promoters will deliver hygiene promotion through an activity that provoke the feeling of comfort by having clean hands. Hygiene promoters will deliver this intervention to up to 5 neighbor households at the time, sharing a story about a family that keeps good hygiene behaviors and therefore are clean, healthy and happy. This story is believed to encourage families to increase handwashing with soap in the household.
  Interventions: Behavioral: Hand hygiene interventions
- Education session for hygiene promotion (No Intervention): Hygiene promoters will deliver regular hygiene promotion activities; an educational message about disease transmission and how handwashing with soap can help protect against disease. This would include teaching participants about the benefits of handwashing with soap, such as reducing diarrhea incidence and preventing cholera.
- Hygiene Promotion Activity - Disgust (Experimental): The activity will be delivered to a group of maximum 5 neighbouring households at the time. Hygiene promoters will use 5 buckets of clean water and place them in front of households. They will then ask a member of one of the households to rinse their hands in the first bucket. Some dirt will come of their hands. Then the participant rinses their hands again in bucket number 2, then 3 and then 4. Before the 5th bucket the participant receives a bar of soap to use when they rinse their hand. When they do the water will have a dirty colour as the dirt comes of their hands. This activity is believed to encourage handwashing with soap.
  Interventions: Behavioral: Hand hygiene interventions
- Hygiene Promotion Activity - Comfort (Experimental): The activity will be delivered to a group of maximum 5 neighbouring households at the time. Hygiene promoters will bring some food oil and ask participants to cover their hands in food oil. They will then ask the participants to cover their hands in turmeric powder. The participants will then be asked to wash their hands with water only. This will have little effect on the cleanliness of their hands. Then participants will be given a bar of soap. The participants will then be asked to wash their hands again. This will leave their hands nice comfortable and clean. They will experience the comfort of clean hands and the activity hope to increase regular handwashing.
  Interventions: Behavioral: Hand hygiene interventions
- Education Hygiene Promotion Activity (No Intervention): Hygiene promoters will deliver regular hygiene promotion activities; an educational message about disease transmission and how handwashing with soap can help protect against disease. This would include teaching participants about the benefits of handwashing with soap, such as reducing diarrhea incidence and preventing cholera.

INTERVENTIONS:
Behavioral: Hand hygiene interventions — Interventions are commonly used physical props for handwashing and commonly used hygiene promotion activities.
  Arms: Bar soap (250gram); Comfort story for hygiene promotion; Hygiene Promotion Activity - Comfort; Hygiene Promotion Activity - Disgust; Mirror (50x30cm); Normal Liquid Soap (250mL); Nurture story for hygiene promotion

SUMMARY:
Understanding how different types of visual prompts and props could impact handwashing practices in humanitarian emergency settings could allow organisations managing camps to deliver hygiene interventions tailored to populations in humanitarian crises. The study aims to test how liquid soap, bar soap and the use of a mirror could impact handwashing behaviours. As such, this research could lead to participants increased handwashing, which should lead to decreased disease transmission of important infectious diseases. With the compliance of NGOs, and the working relationship that will be formed, the results of the research will be shared directly with them. It is likely they will immediately act on any findings.

DETAILED DESCRIPTION:
According to UNICEF, respiratory and diarrheal diseases are the first and second leading causes of deaths among children under-five years of age worldwide. Handwashing has the potential to reduce diarrhoeal disease by almost half and respiratory infections by a quarter. Internally Displaced Persons (IDPs) are especially vulnerable to diarrheal and respiratory diseases, mainly due to overcrowding of settlements and camps and lack of access to WASH facilities. Hygiene programmes delivered in humanitarian crises primarily involve distributing hygiene kits and teaching people about disease transmission. These things are important but are commonly insufficient to lead to behaviour change.

Research in non-emergency settings has shown that the presence of a convenient and desirable handwashing facility may be the factor most likely to determine whether or not people wash their hands. This is particularly relevant to handwashing promotion in IDP camps where it is typically the responsibility of governments or organisations to provide water, sanitation and hygiene (WASH) facilities. Research in non-emergency settings has also shown that using stories and emotional motivators can be a powerful way of changing behaviour, but to date such approaches have not been tried in emergency settings, where they could potentially have a more substantial impact on disease transmission.

Study Aim: To develop and test innovative behaviour change approaches to improve handwashing behaviour among IDPs in Ethiopia.

Study objectives:

1. To conduct a cluster randomised pilot study to assess whether the provision of liquid soap makes handwashing more desirable and more likely to be practiced.
2. To conduct a cluster randomised pilot study to assess whether installing mirrors above the handwashing facility makes handwashing more desirable and more likely to be practiced.
3. To conduct a pilot study of the effect of motivational stories on handwashing behaviour.
4. To conduct a pilot study of the effect of educational activities on handwashing behaviour.

Methodology: The study will be conducted in IDP settlements in Oromia Region. Zones of the camp will be randomised to either receive one of the interventions or to act as a control. If the intervention is successful, the control arm will receive the intervention also. Households will be informed about the research and provide voluntary consent if they wish to participate. Handwashing behaviour will be assessed through structured observation and socio-demographic information will be collected through a survey. Focus groups will be conducted to understand people's perceptions about the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Internally displaces persons living in humanitarian crises settings

Exclusion Criteria:

* Host community

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Structured observation to measure frequency of handwashing, who is washing their hands and whether soap was used. | 4 weeks after implementation
  The primary outcome measure for this study will be observed handwashing at five key critical times (after using the toilet, before preparing food, before eating, before feeding a child and after cleaning a child's faeces). It will also be monitored whether hands are washed with soap or with water only. This will be measured via 3-hour structured observations which is considered to be the gold standard within the sector
Survey on socio-demographics and hand hygiene behaviours | 4 weeks after implementation
  After completing the structured observation, a short survey will be conducted with each household. This will cover family demographics, and information about water, sanitation and hygiene practices. The survey will be administered to the female head of the household. It is estimated that this will take 30 minutes to complete.
Focus group discussions on drivers and barriers to handwashing in the IDP settlement | 1 hour per focus group discussion 6 weeks after implementation
  Focus group discussions will be conducted with recipients in the intervention arms. These will be designed to explore reactions to the interventions and generate reflections on what was liked or disliked about them. The focus group discussions aim to explore what is driving handwashing behaviour, or preventing it in the camps. Two focus group discussions, one with women and one with men, will be conducted in each of the intervention arms. It is estimated that about seven people will participate in each group discussion. Participants will be selected to represent a diverse mix of demographics within the camp and will be individuals that are believed yo contribute most to our learning about hygiene in the local context. The focus group discussions will involve participatory activities using visual prompts or tasks like ranking and scaling. Focus group discussions will be audio recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- London School of Hygiene and Tropical Medecine, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thorseth AH, Heath T, Sisay A, Hamo M, White S. An exploratory pilot study of the effect of modified hygiene kits on handwashing with soap among internally displaced persons in Ethiopia. Confl Health. 2021 May 4;15(1):35. doi: 10.1186/s13031-021-00368-3. PMID 33947443